CLINICAL TRIAL: NCT00650130
Title: DRUID Sub-study: Substance Concentration Ratio/Impairment
Brief Title: Whole Blood-plasma-oral Fluid Ratios of Psychoactive Drugs and Medicines
Status: Completed | Type: Observational
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: University of Helsinki (Other); Ministry of Internal Affairs, Finland (Unknown); European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: KTL 417-7
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-11

CONDITIONS: Driving Under the Influence
Keywords: driving under the influence; psychoactive substances; oral fluid; whole blood; plasma; Ratio of psychoactive substances in whole blood-plasma-oral fluid; Prevalence of psychoactive substances in road traffic
MeSH Terms: conditions — Driving Under the Influence

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — Blood samples and oral fluid are collected for the study. However no DNA detection is done at any stage. The laboratory where samples are analysed do not analyse DNA. DNA is not relevant to this study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: drivers of motorised vehicles suspected of being under the influence of psychoactive drugs

SUMMARY:
The aim of this study is to get new information on the whole blood-plasma-oral fluid ratios of psychoactive drugs which are encountered in traffic.

Samples are taken from drivers suspected of being under the influence of drugs or medicines. The samples are analysed with immunological methods and GC-MS.

Observations from Police and a physician on impairment are combined with the results of the different bodily fluids. Observational evaluations and substance concentrations are compared.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* driver of a motorised vehicle

Exclusion Criteria:

* 17 years or younger
* not the driver of a motorised vehicle

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: drivers of motorised vehicles in general road traffic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
ratio of psychoactive drugs/medicines in whole blood-plasma-saliva and correlation to symptoms of impairment | 1 year

SECONDARY OUTCOMES:
prevalence of psychoactive substances in the general driving population | three years

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Lillsunde, Dr, Principal Investigator — National Public Health Institute, Helsinki, Finland
Locations (1):
- National Public Health Institute, Helsinki, Finland

REFERENCES:
- See also: Official home page of the EU-project — http://www.druid-project.eu